CLINICAL TRIAL: NCT01207908
Title: IGF-1 Therapy and Muscle Function in Duchenne Muscular Dystrophy
Brief Title: Safety and Efficacy Study of IGF-1 in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Ipsen (Industry); Charley's Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-1491
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne Muscular Dystrophy; Insulin like growth factor; 6 minute walk test
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Insulin-Like Growth Factor I; mecasermin; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IGF-1 (Experimental): IGF-1 plus standard steroid treatment
  Interventions: Drug: IGF-1
- Standard steroid treatment alone (No Intervention): Standard daily steroid treatment for DMD

INTERVENTIONS:
Drug: IGF-1 — IGF-1 will be administered once daily by subcutaneous injection every morning with breakfast. Duration 6 months.
  Other Names: Increlex (mecasermin [rDNA origin] injection)
  Arms: IGF-1

SUMMARY:
The purpose of this study is to determine whether IGF-1 therapy improves or preserves muscle function in Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
Detailed Description:

DMD is a progressive degenerative muscle disorder for which there is no current cure. Glucocorticoids (GC) are often used to improve motor function and survival but have significant side effects such as growth failure, weight gain, insulin resistance and osteoporosis. IGF-1 stimulates both the proliferation and differentiation of skeletal muscle cells and is thus important for muscle repair and regeneration. IGF-1 offers potential as a therapeutic agent for DMD as it may improve or preserve motor function and reduce GC side effects such as growth failure and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* DMD diagnosed with mutational testing and/or complete absence of dystrophin on muscle biopsy
* Proximal pelvic girdle weakness (Gower's maneuver, difficulty with arising from floor and going up steps)
* Male
* Age > 5 years of age
* Bone maturation (assess by bone age x-ray): </= 11 years of age
* Daily GC (prednisone or deflazacort) therapy for > 12 months
* Ambulatory
* Informed consent
* Willingness and ability to comply with all protocol requirements and procedures

Exclusion Criteria:

* Current or prior treatment with growth hormone or IGF-1 therapy
* Non-ambulatory
* Pubertal (based on clinical Tanner staging examination)
* Congestive cardiac failure
* History of intracranial hypertension
* Daytime ventilatory dependence (non-invasive or tracheostomy)
* Concomitant therapy - any other medications/supplements that would be considered, in the opinion of the investigators, to affect muscle function, need to have been started 3 months prior to enrollment
* Patients enrolled in other clinical drug trials
* Any physical or mental conditions which may, in the investigators'opinions, render the subject unable to complete the tasks of the study appropriately
* There will be no selection by ethnicity

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meilan Rutter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: Duchenne and Becker Muscular Dystrophy — http://ghr.nlm.nih.gov/condition/duchenne-and-becker-muscular-dystrophy
- See also: Muscular Dystrophy — http://www.nlm.nih.gov/medlineplus/musculardystrophy.html
- See also: Medline — http://www.nlm.nih.gov/medlineplus/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Steroid Treatment Alone: Once daily steroid treatment (Deflazacort or Prednisone) administered orally for DMD.
Period: Overall Study
Arm/Group | IGF-1 | Standard Steroid Treatment Alone
Started | 22 | 22
Completed | 17 | 21
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGF-1 | Standard Steroid Treatment Alone | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.56 (1.28) | 8.70 (1.79) | 8.64 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Difference in 6-Minute Walk Distance Between Groups (Control Minus IGF-1) for Change at 6 Months Versus Baseline
Description: Outcome Measure Data Table shows change of 6-Minute Walk Distance at 6 months versus baseline in each arm. The Statistical Analysis section shows the 6-month difference between the 2 arms (control minus IGF-1).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | IGF-1 | Standard Steroid Treatment Alone
Number analyzed (Participants) | 17 | 21
meters | 3.4 (32.4) | -5.1 (50.2)
Statistical Analysis 1: Comparison: IGF-1 vs Standard Steroid Treatment Alone; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-37.1 to 20.1]

2. Secondary Outcome: Difference in Height Velocity Between Groups (Control Minus IGF-1) for Change at 6 Months Versus Baseline
Description: Outcome Measure Data Table shows change of height velocity at 6 months versus baseline in each arm. The Statistical Analysis section shows the 6-month difference between the 2 arms (control minus IGF-1).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | IGF-1 | Standard Steroid Treatment Alone
Number analyzed (Participants) | 17 | 21
cm/year | 2.60 (1.64) | -0.06 (1.69)
Statistical Analysis 1: Comparison: IGF-1 vs Standard Steroid Treatment Alone; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -2.66, 95% CI 2-sided [-3.78 to -1.55]

3. Secondary Outcome: Difference in North Star Ambulatory Assessment (NSAA) Score Between Groups (Control Minus IGF-1) for Change at 6 Months Versus Baseline
Description: Outcome Measure Data Table shows change of North Star Ambulatory Assessment (NSAA) score at 6 months versus baseline in each arm. The Statistical Analysis section shows the 6-month difference between the 2 arms (control minus IGF-1).
  The NSAA is a 17-item scale that grades performance of various functional skills on a scale from 0 (unable), 1 (complete independently but with modifications), and 2 (complete without compensation).
  The range of NSAA score is from 0 to 34. The higher score indicates better motor function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGF-1 | Standard Steroid Treatment Alone
Number analyzed (Participants) | 17 | 21
score on a scale | -0.94 (2.41) | -0.4 (3.0)
Statistical Analysis 1: Comparison: IGF-1 vs Standard Steroid Treatment Alone; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-1.26 to 2.38]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | IGF-1 | Standard Steroid Treatment Alone
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 20/22 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGF-1 (N=22) | Standard Steroid Treatment Alone (N=22)
Intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | IGF-1 (N=22) | Standard Steroid Treatment Alone (N=22)
Headache (Nervous system disorders) | 11 | 9
Nausea and vomiting (Gastrointestinal disorders) | 7 | 5
seizure (Nervous system disorders) | 0 | 1
papilledema (Nervous system disorders) | 1 | 0
stinging at injection site (Skin and subcutaneous tissue disorders) | 3 | 0/0 — The control group was not considered at risk for this adverse event because they did not receive any injections. Therefore the denominator here is zero.
fever (General disorders) | 2 | 3
rash and skin welt (Skin and subcutaneous tissue disorders) | 3 | 1
lipohypertrophy (Musculoskeletal and connective tissue disorders) | 4 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Finger injury (Musculoskeletal and connective tissue disorders) | 1 | 1
Leg injury (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Finger infection (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Arm weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg numbness (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Small sample size and short duration, Open-label study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes